CLINICAL TRIAL: NCT04076176
Title: The Effects Of Casein Glycomacropeptide On Metabolic Control And General Health Status In Children And Adults With PKU: A Randomised Crossover Trial
Brief Title: The Effects of CGMP in Children and Adults With PKU
Acronym: ELEMENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Collaborators: Arla Foods (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MCT-CGMP-2017-05-23; 239520 (Other: IRAS); 19/NW/0032 (Other: HRA)
Record Dates: First submitted 2019-05-30; First posted 2019-09-03 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Phenylketonurias
Keywords: Phenylketonuria; PKU; Child; Adult; GMP; Glycomacropeptide
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-amino Acids (Active Comparator): The specific amount and timing of L-amino acid consumption will be at the instruction of a dietitian following a review of the individual patient's dietary needs.
  Consumption period: 12 weeks.
  Interventions: Dietary Supplement: L-amino acid protein substitute
- PKU Sphere (Experimental): The specific amount and timing of PKU sphere consumption will be at the instruction of a dietitian following a review of the individual patient's dietary needs.
  Consumption period: 12 weeks.
  Interventions: Dietary Supplement: CGMP protein substitute

INTERVENTIONS:
Dietary Supplement: CGMP protein substitute — PKU sphere is a powdered, low phenylalanine protein substitute, containing a balanced mix of casein glycomacropeptide (CGMP) isolate, essential and non-essential amino acids, carbohydrate, vitamins, minerals, trace elements and the omega-3 long chain polyunsaturated fatty acid (LCP); docosahexaenoic acid.
  Other Names: PKU Sphere
  Arms: PKU Sphere
Dietary Supplement: L-amino acid protein substitute — Patient may choose from a list of products, specified in the protocol, that are nutritionally comparable to PKU Sphere.
  Arms: L-amino Acids

SUMMARY:
Randomised controlled trial with a crossover design. For early and continuously treated patients with phenylketonuria (PKU) that are adherent. Two 12-week periods where patients consume either casein glycomacropeptide (CGMP) based protein substitute or a free amino acid (AA) based protein substitute. 4 week wash out period in between. The protein substitutes will be consumed daily together with the patient's regular low protein diet.

DETAILED DESCRIPTION:
The study is a randomised controlled trial with a crossover design conducted at several international study centres.

The study population is early and continuously treated patients with PKU that are adhering to their prescribed diet.

The participants will be given both a CGMP based protein substitute and a free AA based protein substitute as their main protein source on two different 12-week periods in a crossover design. The two periods will be separated by a 4 week wash out period.

The protein substitutes will be consumed daily together with the patient's regular low protein diet during the intervention periods.

Primary Objective The primary objective of the study is to investigate the effects of a CGMP based formula compared to an AA based formula upon mean plasma Phe levels after 12 weeks of daily intake in patients with PKU.

Secondary Objectives The secondary objectives of the study are to investigate if a CGMP based formula compared to an AA based formula in PKU patients provides any long-term health benefits concerning gut health, inflammation, oxidative stress and product acceptability.

ELIGIBILITY:
Inclusion Criteria:

* PKU patient diagnosed on newborn screening (NBS).
* > 50% of protein intake from protein substitutes.
* (CHILDREN) Dietary intake of ≤ 1000 mg Phe from natural protein or ≤20 g natural protein inclusive of fruit and vegetables per day.
* (ADULTS) Dietary intake of ≤ 1500 mg Phe from natural protein or ≤ 30 g natural protein inclusive of fruit and vegetables per day.
* (CHILDREN) Three out of the last four consecutive Phe measurements within the target range (≤360 µmol/L in patients aged 4-12 years).
* (ADULTS) Two out of the last four consecutive Phe measurements within the target range (≤600 µmol/L for adults).
* Male or female aged 4-12 years or 18 years and over.
* Early and continuously treated. Adherent to their prescribed PKU diet consisting of a protein-restricted diet and free AA based protein substitute.
* Otherwise in good general health as evidenced by medical history.
* Able to provide written informed consent (patient or parent/guardian).
* Able to comply with the study protocol and take study product according to the opinion of the PI.
* Protein substitute intake provided by L-amino acid supplements only.
* (ADULTS) No studies have been done in pregnant women. To ensure patients safety, female patients of childbearing potential must have a negative pregnancy test prior to completing the screening procedures.
* (ADULTS) All female patients of childbearing potential and sexually mature males should be willing to use a medically accepted method of contraception throughout the study.
* Successful 3-day PKU Sphere taste test.

Exclusion Criteria:

* Concomitant diseases / disorders such as but not limited to renal or gut disease / disorders and diabetes.
* Currently or previously treated with tetrahydrobiopterin (BH4), pegylated recombinant phenylalanine ammonia lyase (PEG PAL), large neutral amino acids.
* Previous intake of CGMP for more than four consecutive weeks.
* Having a current infection.
* Known soya, milk or fish allergies / intolerance.
* Patients who are currently participating in, plan to participate in, or have participated in an interventional investigational drug, food or medical device trial within 30 days prior to screening visit.
* Where applicable, patients not covered by Health Insurance System and/or not in compliance with the recommendations of National Law in force.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change in overnight fasting plasma Phe | Measured at days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5)
  Overnight fasting plasma phenylalanine level (μmol/l)
Change in overnight fasting plasma Tyr | Measured at days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5)
  Overnight fasting plasma tyrosine level (μmol/l)
Change in overnight fasting blood Phe | Measured twice per week up to 32 weeks
  Overnight fasting blood phenylalanine level (μmol/l) using blood spots
Change in overnight fasting blood Tyr | Measured twice per week up to 32 weeks
  Overnight fasting blood tyrosine level (μmol/l) using blood spots

SECONDARY OUTCOMES:
Change in gut health: PedsQL Gastrointestinal Symptoms Scales, Version 3.0 | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Five point frequency scale for each question: Never (0), Almost Never (1), Sometimes (2), Often (3), Almost Always (4).
Change in gut health: Stool pH for reducing sugars | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  From stool sample. To rule out carbohydrate intolerance as a cause of any irritable bowel syndrome symptoms
Change in gut health: Stool calprotectin | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  From stool sample
Change in gut health: Short chain fatty acids | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  From stool sample
Change in gut health: Immunoglobulin A | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  From stool sample
Change in gut health: Bristol stool form scale | Completed for 7 days prior to days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Bristol stool form scale:
  * Type 1: Separate hard lumps, like nuts (hard to pass)
  * Type 2: Sausage-shaped, but lumpy
  * Type 3: Like a sausage but with cracks on its surface
  * Type 4: Like a sausage or snake, smooth and soft
  * Type 5: Soft blobs with clear cut edges (easy to pass)
  * Type 6: Fluffy pieces with ragged edges, a mushy stool
  * Type 7: Watery, no solid pieces, entirely liquid
Change in gut health: 3 day weighed diet diary | Completed for 3 days prior to days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  3 day weighed diet diary
Change in anthropometric measurements: weight | Days -31 (visit 1), 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Weight (kg)
Change in anthropometric measurements: height | Days -31 (visit 1), 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Height (cm)
Change in Albumin | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Following overnight fasting
Change in Pre-albumin | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Following overnight fasting
Change in Transferrin | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Following overnight fasting
Change in Retinol-binding protein | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Following overnight fasting
Change in Glucose | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Following overnight fasting
Change in Haemoglobin A1C | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Following overnight fasting
Change in IGF-1 | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Following overnight fasting
Change in C-peptide | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Following overnight fasting
Change in Short chain fatty acids | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Following overnight fasting
Change insulin production | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Following overnight fasting
Change in alanine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in arginine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in asparagine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in citrulline | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in cystine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in glutamate | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in glutamine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in glycine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in histidine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in isoleucine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in leucine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in lysine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in methionine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in proline | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in ornithine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in phenylalanine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in serine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in taurine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in threonine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in tryptophan | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in tyrosine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in valine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Total plasma amino acids following overnight fasting
Change in renal biomarkers: Serum cystatin C | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Blood sample following overnight fasting
Change in renal biomarkers: Serum creatinine | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Blood sample following overnight fasting
Change in renal biomarkers: Blood urea nitrogen | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Blood sample following overnight fasting
Change in Adiponectin | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Following overnight fasting. An anti-inflammatory marker and related with both adipose tissue and insulin sensitivity
Change in C-reactive protein (high sensitivity measurement) | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Following overnight fasting
Change in Serum myeloid-related protein | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Following overnight fasting
Change in Soluble Interleukin 2 Receptor | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Following overnight fasting
Change in Inflammatory cytokine panel | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Following overnight fasting
Change in oxidative stress: White cells glutathione (GSH) | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Following overnight fasting
Change in oxidative stress: Plasma thiobarbituric acid-reactive species (TBAR) | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Following overnight fasting
Change in oxidative stress:Total antioxidant reactivity (TAR) | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5).
  Following overnight fasting
Change in patient opinion of acceptability of the product | Days 84 (visit 3) and 196 (visit 5)
  Product acceptability Likert scale:
  * I loved it (5 - best)
  * I liked it (4)
  * I neither liked nor disliked it (3)
  * I didn't like it (2)
  * I really didn't like it (1 - worst)
Change in hunger | Days 0 (visit 2), 84 (visit 3), 112 (visit 4) and 196 (visit 5)
  Measuring hunger in primary school children Likert scale:
  * I am really hungry! My belly feels very empty and is rumbling! (1 - worst)
  * I am quite hungry and my belly feels a little empty. (2)
  * I feel just right, not too hungry and not too full. (3)
  * I am quite full, but there is still a little room in my belly. (4)
  * I am not hungry at all! My belly feels very full and I cannot eat any more food! (5 - best)

CONTACTS AND LOCATIONS:
Overall Officials: Anita MacDonald, Principal Investigator — Birmingham Women's and Children's NHS Foundation Trust
Locations (3):
- Rigshospitalet, Copenhagen, Denmark
- United Kingdom (2):
  - Bristol Royal Hospital for Children, Bristol, Avon
  - Birmingham Children's Hospital, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pinto A, Daly A, Newby C, Robotham A, Heales S, Eaton S, Aitkenhead H, Gilmour K, Jackson R, Ashmore C, Evans S, Rocha JC, Ilgaz F, Hickson M, MacDonald A. The effects of casein glycomacropeptide on general health status in children with PKU: A randomized crossover trial. Mol Genet Metab. 2024 Dec;143(4):108607. doi: 10.1016/j.ymgme.2024.108607. Epub 2024 Nov 4. PMID 39579672